CLINICAL TRIAL: NCT02217319
Title: Does a Sevoflurane Preconditioning Have Cardioprotective Properties in Noncardiac Thoracic Surgery?
Brief Title: Cardioprotection by Sevoflurane Preconditioning in Noncardiac Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSK005
Record Dates: First submitted 2014-08-08; First posted 2014-08-15 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: High Sensitive Troponin T Release
Keywords: Volatile Anesthetic; Cardioprotection; Lung surgery; non cardiac surgery
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Active Comparator): Patients receive Sevoflurane 1 MAC (minimal alveolar concentration) after induction of anesthesia with propofol, remifentanil and atracurium for 30 minutes as preconditioning.
  Interventions: Drug: Sevoflurane
- TIVA (Placebo Comparator): Patients received the standard total intravenous anesthesia (TIVA) with propofol, remifentanil and atracurium.
  Interventions: Drug: TIVA

INTERVENTIONS:
Drug: Sevoflurane — Anaesthesia is induced (1-2 mg/kg) and maintained (5-7 mg/kg/h) with propofol and remifentanil (1 µg/kg and 0,2-0,4 µg/kg/min). After induction of anesthesia the propofol infusion is stopped and patients receive 1 MAC Sevoflurane over 30 min. Then the propofol infusion is restarted and Sevoflurane is washed out.
  Arms: Sevoflurane
Drug: TIVA — Anaesthesia is induced (1-2 mg/kg) and maintained (5-7 mg/kg/h) with propofol and remifentanil (1 µg/kg and 0,2-0,4 µg/kg/min).
  Other Names: Placebo; Controll
  Arms: TIVA

SUMMARY:
It has been shown that the use of volatile anaesthetics, that are usually used to perform a general anesthesia, have cardioprotective properties. This has been shown in animal studies and in patients that underwent cardiac surgery. The aim of our study is to examine if Sevoflurane, a volatile anaesthetic, has this properties in patients undergoing lung surgery.

ELIGIBILITY:
Inclusion Criteria:

* Lung surgery
* ASA (American Society of Anesthesiologists) physical status 1-3

Exclusion Criteria:

* Disposition for malignant hyperthermia
* Medication with ß-blocking drugs
* Use of clonidin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Troponin T | change of Troponin T levels preoperative and postoperative up to 40 hours after surgery
  assessing a change in high sensitive Troponin T (5th generation) Level before and at six time points after surgery (right after surgery, every 8 hours up to 40 hours after surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Horst Schmidt Klinik, Wiesbaden, Germany